CLINICAL TRIAL: NCT06116461
Title: Nivolumab Dose Optimization in Patients With a Complete, Partial or Stable Response
Acronym: NIVOPTIMIZE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, S. L. W. (Stijn) Koolen, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL77343.078.21
Record Dates: First submitted 2023-10-04; First posted 2023-11-03 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Patients in the experimental arm receive three reduced nivolumab doses of 240 mg Q4W
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Participants receive three reduced doses of 240 mg every four weeks

SUMMARY:
Patients with advanced melanoma are, amongst others, currently treated with nivolumab monotherapy or with nivolumab and ipilimumab followed by nivolumab. Even though registration studies administered nivolumab in a 3 mg/kg 2 weekly scheme, currently, nivolumab monotherapy is either administered in a 240 mg 2-weekly scheme or in a 6 mg/kg or 480 mg 4-weekly scheme. With the current dosing regimen, steady-state is achieved after approximately 5 to 6 months, whereas a tumour response is usually observed earlier in patients with metastatic melanoma. Moreover, PD-1 receptor occupancy is almost saturated above doses of 0.3 mg/kg, or at nivolumab serum levels of 10 mg/L, which is a concentration that is achieved after one treatment cycle. In melanoma patients, the additional probability on response in patients treated with 3 mg/kg compared to 1 mg/kg seems limited. PFS and OS for 3 mg/kg were not superior to 1 mg/kg. Therefore, in this study, our aim is to investigate nivolumab trough levels and pharmacokinetic parameters after 3 reduced nivolumab doses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Advanced or metastatic melanoma
* Current treatment with nivolumab for advanced or metastatic melanoma, in a 6 mg/kg or 480 mg, 4 weekly scheme
* Documented confirmed and ongoing CR, PR or SD according to RECIST v1.1
* On treatment for at least 6 months

Exclusion Criteria:

* Unable to draw blood for study purposes
* Patients willing to participate or already included in the SAFE-STOP trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Difference between the nivolumab mean trough level after 3 reduced doses (240 mg every 4 weeks) and after the first dose of 6 mg/kg or 480 mg. | Through study completion, an average of four months
  Difference between the nivolumab mean trough level after 3 reduced doses (240 mg every 4 weeks) and after the first dose of 6 mg/kg or 480 mg.

SECONDARY OUTCOMES:
- PD-1 receptor occupancy in PBMCs, measured 4 weeks after 3 reduced nivolumab doses | Through study completion, an average of four months
  - PD-1 receptor occupancy in PBMCs, measured 4 weeks after 3 reduced nivolumab doses
Grade ≥3 adverse events (CTCAE) during reduced doses | Through study completion, an average of four months
  Grade ≥3 adverse events (CTCAE) during reduced doses
Number of patients with new PD during 3 reduced doses | Through study completion, an average of four months
  Number of patients with new PD during 3 reduced doses

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Pending, Netherlands

IPD SHARING:
Plan to Share IPD: No